CLINICAL TRIAL: NCT03107234
Title: Involvement of the Inositol-trisphosphate Receptor in Invasive or Migratory-type Breast Cancers
Acronym: CarcIno
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0007
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Inosine Triphosphatase
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with breast cancer requiring surgery to
  Interventions: Other: Assess the level of expression of IP3R3 in cancerous tissues and healthy tissues

INTERVENTIONS:
Other: Assess the level of expression of IP3R3 in cancerous tissues and healthy tissues — Assess the level of expression of IP3R3 in cancerous tissues and healthy tissues

SUMMARY:
Breast cancer is the leading cause of female cancer and female death by cancer in France. Despite the improvement in early detection and therapeutic arsenal, the mortality of this cancer remains high with 11 886 deaths estimated in 2012. Breast cancer is most often a carcinoma born from the lobular or ductal epithelium and is classified In two main categories: non invasive and invasive. Invasive breast cancers account for 75% of the cases. They are usually ductal (75%) and more rarely lobular (25%). The cancer cells are then no longer circumscribed to the galactophoric canals or glands but have invaded neighboring tissues. If they are not treated in time, these cancers can then spread: the cancerous cells will then migrate either by the lymphatic vessels to reach the neighboring ganglia or through the blood vessels to give metastases in other tissues In the liver, lungs and bones). The mortality associated with breast cancer is not due to the growth of the primary tumor but rather to the occurrence of metastases. The study of the mechanisms leading to metastatic invasion (i.e. migration and invasion) is therefore of considerable importance. The development of metastases depends on the acquisition by the cancer cells of various capacities including that of being able to migrate, involving a remodeling of the cytoskeleton highly dependent on the intracellular calcium (Ca2 +) concentration. Several types of signals are able to induce mobilization of Ca2 + from the extracellular medium or endoplasmic reticulum (ER) reserves. At the intracellular level, some of these signals are generated by inositol (1,4,5) -trisphosphate (IP3) from the activation of G protein-coupled receptors or certain receptors with tyrosine kinase activity. Has been shown that the expression, activity and regulation of IP3R receptors (IP3Rs) are involved in the cancerous processes of many tissues, in particular in the phenomena of proliferation of breast cancer cells. Overall, altered expression and / or activity of IP3Rs can be used for the survival, growth, proliferation and migration of cancer cells.

In the laboratory, the investigator showed that regulation of the expression of subtype 3 (IP3R3) by 17β-estradiol (E2) is involved in the growth of the human mammary cancer line MCF-7. E2 triggers the release of Ca2 + in an IP3-dependent mechanism, while prolonged exposure to E2 leads to an increase in the expression of IP3R3. At the same time, the reduction in the expression of IP3R3 cancels the proliferative effect of E2 on MCF-7 cells. More recently, the investigator has established that IP3R3 regulates the proliferation of cells of the human MCF-7 mammary cancer cell line via a molecular and functional interaction with the Ca2 + -dependent BKCa potassium channel. The determination of IP3Rs, including subtype 3, as a mediator / marker of breast carcinogenesis appears to be a major clinical issue.

ELIGIBILITY:
Inclusion Criteria:

* CCI / CLI to be operated
* Grade SBR 1, 2 or 3
* Undifferentiated RE / PR status
* HER2 status undifferentiated
* Ki 67 indifferent
* Metastatic or not
* ADP axillary invaded or not
* Major Patients

Exclusion Criteria:

* CIC / CIL
* Males

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with breast cancer requiring surgery to
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-07-17 (Estimated); Study Completion 2018-07-17 (Estimated)

PRIMARY OUTCOMES:
Level of expression of IP3R3 defined by an immunohistochemical score | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France